CLINICAL TRIAL: NCT00500331
Title: A Double-blind, Randomized 12-week Study to Evaluate the Safety and Efficacy of GSK189075 Tablets vs Pioglitazone in Treatment Naive Subjects With Type 2 Diabetes Mellitus
Brief Title: Dose-Ranging Study in Treatment Naive Type 2 Diabetes Mellitus(T2DM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KG2105255
Record Dates: First submitted 2007-01-24; First posted 2007-07-12 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Pioglitazone; HbA1c; Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): GSK189075
  Interventions: Drug: GSK189075
- Arm 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- Arm 3 (Other): pioglitazone (active control)
  Interventions: Drug: pioglitazone

INTERVENTIONS:
Drug: GSK189075 — Experimental Drug
  Arms: Arm 1
Drug: pioglitazone — Active Control
  Arms: Arm 3
Other: Placebo — Placebo Comparator
  Arms: Arm 2

SUMMARY:
This is a dose-ranging study that will evaluate the efficacy, safety and tolerability of a range of doses of investigational product and pioglitazone, compared to placebo, administered as monotherapy over 12 weeks in treatment naive patients with T2DM

ELIGIBILITY:
Inclusion criteria:

* Subjects with a documented diagnosis of T2DM and have an HbA1c level at Visit 1 of ≥7.0% and ≤9.5% as measured by a central laboratory. Subjects with HbA1c <7.5% must have a fasting fingerstick glucose ≥7 mmol/L (126 mg/dL) at Week 0 prior to randomization.
* Subjects who are treatment-naïve and have not taken insulin, or any oral or injectable anti-diabetic medication in the past 3 months and have not taken a glucose lowering agent for ≥4 weeks at any time in the past, or Subjects who are newly diagnosed and treated with diet and exercise for a minimum of 6 weeks
* Subjects who are 18 to 70 years of age inclusive at the time of Screening.
* Females of non-childbearing and childbearing potential are eligible to participate as follows:

  * Women of childbearing potential must be willing to use one of the following contraception methods: intrauterine device, condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent for at least 30 days prior to the start of study medication, throughout the study and the follow-up visit. Note: use of oral contraceptives is not permitted.
  * Women of non-child bearing potential are defined as follows: females regardless of age, with functioning ovaries and who have a current documented tubal ligation [Hatcher, 2004] bilateral oophorectomy or total hysterectomy, or females who are post-menopausal).

(Post-menopausal is defined as after one year without menses with an appropriate clinical profile, e.g. age appropriate, >45 years, in the absence of hormone replacement therapy. In addition to the above criteria, if the post-menopausal status is still questionable, a blood sample should be drawn for simultaneous measurement of follicle stimulating hormone and estradiol; values considered to confirm the post-menopausal state are respectively: FSH >40 MIU/mL and estradiol <40pg/mL (<140 pmol/L)).

* Informed Consent: a signed and dated written consent must be obtained from the subject before any procedures are performed.

Exclusion Criteria:

* Metabolic Disease

  * Diagnosis of Type 1 diabetes mellitus.
  * History of ketoacidosis which has required hospitalization.
  * Thyroid disorder [TSH below the lower limit of the reference range (LLRR) of 0.4mIU/L or above the upper limit of the reference range (ULRR) of >5.5 mIU/L at Screening]. Hypothyroidism treated with the same dose and regimen of thyroid hormone replacement for at least 3 months prior to Screening is allowed.
  * BMI of <22 or >43 kg/m2.
  * Significant weight gain or loss (as defined as >5% of total body weight) in the 3 months prior to Screening.
* Diabetic Medication

  * Has taken insulin or any oral or injectable anti-diabetic medication ≥4 weeks at any time prior to screening.
  * Has taken insulin or any oral or injectable anti-diabetic medication within 3 months of screening.
* Cardiovascular Disease

  * Recent history or presence of clinically significant acute cardiovascular disease including:

    1. Documented myocardial infarction in the 6 months prior to Screening.
    2. Coronary revascularization including percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG) surgery either planned and/or occurred in the 6 months prior to Screening.
    3. Unstable angina in the 6 months prior to Screening.
    4. Clinically significant supraventricular arrhythmias requiring medical therapy, or history of nonsustained or sustained ventricular tachycardia. Symptomatic valvular heart disease or valvular heart disease requiring therapy other than endocarditis prophylaxis.
    5. Congestive heart failure (CHF, New York Heart Association (NYHA) Class II to IV) requiring pharmacologic treatment. NYHA Class I may be included in accordance with the local prescribing information for pioglitazone.
    6. Blood pressure (BP) >150/100mmHg. If a subject is receiving permitted antihypertensive therapy, then they must be on stable dose(s) of therapy for at least 4 weeks prior to Screening.
    7. Has a QTc interval (Bazett's) ≥450msec at Screening on a single ECG or an average value from 3 ECGs taken 5 minutes apart (on local reading of ECG).
    8. Other clinically significant ECG abnormalities which, in the opinion of the investigator, may affect the interpretation of efficacy and safety data, or which otherwise contraindicates participation in a clinical trial with a new chemical entity.
  * Fasting triglycerides ≥400mg/dL (4.56mmol/L) at Screening. If a subject is receiving permitted lipid-lowering therapy, then they must be on a stable dose(s) of therapy for at least 6 weeks prior to Screening. Niacin and bile acid sequestrants are prohibited.
* Hepatic Disease

Has a diagnosis of active hepatitis (hepatitis B surface antigen or hepatitis C antibody), or clinically significant hepatic enzyme elevation including:

Any one of the following enzymes greater than 2 times the upper limit of the reference range (ULRR) value at Screening.

* alanine transaminase (ALT).
* aspartate transaminase (AST).
* alkaline phosphatase (AP). Has a total bilirubin level that is >1.5 times the ULRR at Screening with the exception of suspected or confirmed Gilbert's disease.

  * Pancreatic Disease
* Secondary causes of diabetes:
* history of chronic or acute pancreatitis

  * Renal Disease
* Significant renal disease at Screening as manifested by:

Glomerular filtration rate (GFR) <60mL/min (as estimated from serum creatinine at Visit 1 and demographic data using the MDRD equation).For the MDRD equation, please refer to the study procedures manual.

Proteinuria of ≥1+ by urinary dipstick

* Recurrent genitourinary tract infections defined as ≥2 episodes of complicated or uncomplicated cystitis or pyelonephritis in the 6 months prior to Screening
* A positive qualitative urinary dipstick for leukocytes, red blood cells (RBC) or nitrites at Screening.

  * Concurrent Disease
* Has any concurrent condition or any clinically significant abnormality identified on the screening physical examination, laboratory tests (including blood electrolytes), electrocardiogram, including pulmonary, neurological or inflammatory diseases, which, in the opinion of the investigator, may affect the interpretation of efficacy and safety data, or which otherwise contraindicates participation in a clinical trial with a new chemical entity
* History of significant co-morbid diseases active in the 6 months prior to Screening (e.g., cholecystitis, acute pancreatitis, gastrointestinal disease, chronic diarrhea, etc.)
* Has a history of malignancy within the past five years [other than superficial squamous cell carcinoma which is non-invasive on pathology or basal cell carcinoma which is successfully treated with local excision] and cervical cancer in situ treated definitively at least 6 months prior to Screening

  * Concurrent Medication
* Is currently taking or has taken any of the following medications in the 8 weeks prior to Screening:

  1. Digoxin
  2. Warfarin and other oral anticoagulants (aspirin and non-steroidal anti-inflammatory drugs are permitted)
  3. Bile acid sequestrants
  4. Niacin (excluding routine vitamin supplementation)
  5. Antiobesity agents (including fat absorption blocking agents)
  6. Oral or injectable corticosteroids (inhaled and intranasal corticosteroids are permitted)
  7. Loop diuretics
  8. Monoamine oxidase inhibitors and tricyclic amines
  9. Antiretroviral drugs
  10. St John's Wort
  11. Oral chromium

      * Pregnancy & Breast Feeding
* Is currently lactating or pregnant

  * Other
* Current smoker who is unable to abstain from smoking while in the clinic at each visit
* Has a history of alcohol or substance abuse within the past year at Screening or alcohol or substance abuse during treatment, as determined by the investigator:
* Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* Has an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males) or an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half-pint of beer or 1 measure of spirits or 1 glass of wine
* Has participated in any study with an investigational or marketed drug in the 3 months prior to Screening
* In the opinion of the investigator has a risk of non-compliance with study procedures, or cannot read, understand, or complete study related materials, particularly the informed consent
* Known allergy to any of the tablet excipients, or history of drug or other allergy, which, in the opinion of the responsible study physician

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2007-01-23 (Actual); Primary Completion 2008-02-14 (Actual); Study Completion 2008-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (107):
- United States (12):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Saint Cloud, Florida
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Oxon Hill, Maryland
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Canal Fulton, Ohio
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Burke, Virginia
- Argentina (9):
  - GSK Investigational Site, Buenos Aries, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Quilmes
  - GSK Investigational Site, San Miguel de Tucumán
- Bulgaria (4):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- GSK Investigational Site, San José, Costa Rica
- Czechia (10):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Cheb
  - GSK Investigational Site, České Budějovice
  - GSK Investigational Site, Havirov - Soumbrak
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Semily
  - GSK Investigational Site, Šumperk
  - GSK Investigational Site, Ústí nad Labem
  - GSK Investigational Site, Znojmo
- Germany (15):
  - GSK Investigational Site, Bammental, Baden-Wurttemberg
  - GSK Investigational Site, Kippenheim, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Haag, Bavaria
  - GSK Investigational Site, Höhenkirchen-Siegertsbrunn, Bavaria
  - GSK Investigational Site, Lampertheim, Hesse
  - GSK Investigational Site, Damme, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Hildesheim, Lower Saxony
  - GSK Investigational Site, Bergkamen, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Speyer, Rhineland-Palatinate
  - GSK Investigational Site, Berlin
- Hungary (13):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Érd
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Mosonmagyaróvár
  - GSK Investigational Site, Nyirtegyhaza
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Szentes
  - GSK Investigational Site, Szigetvár
  - GSK Investigational Site, Szombathely
  - GSK Investigational Site, Veszprém
  - GSK Investigational Site, Zalaegerszeg
- India (5):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
- Latvia (5):
  - GSK Investigational Site, Jelgava
  - GSK Investigational Site, Limbaži
  - GSK Investigational Site, Riga
  - GSK Investigational Site, Talsi
  - GSK Investigational Site, Tukums
- Lithuania (2):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Vilnius
- Mexico (5):
  - GSK Investigational Site, Tijuana, Baja California Norte
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, México, State of Mexico
  - GSK Investigational Site, Durango
  - GSK Investigational Site, México
- New Zealand (3):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Rotorua
- GSK Investigational Site, Lima, Peru
- Poland (6):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Grudziądz
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Porąbka
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Wroclaw
- GSK Investigational Site, Ponce, Puerto Rico
- Romania (4):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Iași
- Russia (5):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Tyumen
  - GSK Investigational Site, Ufa
- South Africa (5):
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Gauteng
  - GSK Investigational Site, Orangegrove, Linksfield West
  - GSK Investigational Site, Parow
  - GSK Investigational Site, Roodepoort

REFERENCES:
- [Derived] Sykes AP, O'Connor-Semmes R, Dobbins R, Dorey DJ, Lorimer JD, Walker S, Wilkison WO, Kler L. Randomized trial showing efficacy and safety of twice-daily remogliflozin etabonate for the treatment of type 2 diabetes. Diabetes Obes Metab. 2015 Jan;17(1):94-7. doi: 10.1111/dom.12391. Epub 2014 Nov 3. PMID 25223369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 121 centers of which 95 randomized participants, in 18 countries (9 European, 8 International, and the United States) from 23 January 2007 to 14 February 2008.
Pre-assignment Details: The Screening period was of 2 weeks. A glucose meter and detailed instructions for use were provided to all participants at the Screening visit for self- monitoring of fasting blood glucose levels and a Daily Glucose Monitoring Log for recording blood glucose information. Dietary and exercise advice was provided at randomization.
Groups:
- Placebo: Eligible participants received matching placebo, orally, twice daily before breakfast and dinner for 12 weeks.
- GSK189075 50 mg: Eligible participants received GSK189075 50 milligram (mg) tablets, orally, twice daily before breakfast and dinner for 12 weeks.
- GSK189075 100 mg: Eligible participants received GSK189075 100 mg tablets, orally, twice daily before breakfast and dinner for 12 weeks.
- GSK189075 250 mg: Eligible participants received GSK189075 250 mg tablets, orally, twice daily before breakfast and dinner for 12 weeks.
- GSK189075 500 mg: Eligible participants received GSK189075 500 mg tablets, orally, twice daily before breakfast and dinner for 12 weeks.
- GSK189075 1000 mg: Eligible participants received GSK189075 1000 mg tablets, orally, twice daily before breakfast and dinner for 12 weeks.
- Pioglitazone 30 mg: Eligible participants received Pioglitazone 30 mg tablets, orally, once daily before breakfast for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Started | 48 | 47 | 48 | 48 | 48 | 47 | 48
Completed | 33 | 42 | 43 | 38 | 44 | 42 | 46
Not Completed | 15 | 5 | 5 | 10 | 4 | 5 | 2
Not completed — Adverse Event | 0 | 2 | 0 | 1 | 2 | 2 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 2 | 1 | 0 | 0
Not completed — Protocol Violation | 3 | 1 | 1 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 0 | 1 | 5 | 0 | 1 | 1
Not completed — Lack of Efficacy | 3 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Liver function test abnormality | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Increased serum creatinine from Baseline | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Didn't return for continuation of study | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Exclusion citeria not met on Visit 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor decided to withdraw participant | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant was randomized by mistake | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Diabetologist nurse in the study | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — State ban of biological samples export | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol violated | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK189075 50 mg: Eligible participants received GSK189075 50 mg tablets, orally, twice daily before breakfast and dinner for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg | Total
Number analyzed (Participants) | 48 | 47 | 48 | 48 | 48 | 47 | 48 | 334
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.9 (9.67) | 54.3 (9.04) | 56.0 (8.11) | 55.7 (9.46) | 54.6 (9.33) | 52.4 (9.03) | 54.5 (9.45) | 54.8 (9.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 17 | 19 | 20 | 20 | 24 | 141
  Male | 30 | 24 | 31 | 29 | 28 | 27 | 24 | 193
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 4 | 3 | 0 | 3 | 4 | 19
  Asian | 1 | 2 | 3 | 1 | 2 | 1 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 4
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 41 | 37 | 36 | 41 | 42 | 40 | 39 | 276
  More than one race | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 5
  Unknown or Not Reported | 3 | 2 | 2 | 2 | 3 | 2 | 2 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Week 0) in Glycosylated Hemoglobin (HbA1c) (%) at Week 12
Description: Fasted blood samples for HbA1c were collected at Baseline and Week 12. Participants were required to fast for at least 8 hours prior to laboratory samples and were told not to take the morning dose of study medication on these visit days and to refrain from eating until instructed to do so by study personnel in the clinic. When the participant had not fasted, the participant was rescheduled to return to the clinic to have a fasted sample taken. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. Only those participants with a value at Baseline and at Week 12 (after Last Observation Carried Forward [LOCF]) were used for this analysis. Adjusted mean is presented as least square mean.
Time Frame: Baseline (Week 0) and Week 12
Population: Intent to Treat (ITT) Population with LOCF comprised of all randomized participants who received at least one dose of randomized study medication, had a Baseline assessment and had at least one corresponding on-therapy (scheduled or unscheduled) efficacy assessment. One extreme outlier participant had withdrawn from Placebo arm (lack of efficacy).
Measure: Least Squares Mean (Standard Error); unit: Percentage of hemoglobin
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 43 | 45 | 43 | 44 | 47 | 45 | 47
Percentage of hemoglobin | -0.31 (0.107) | -1.04 (0.105) | -0.96 (0.107) | -1.05 (0.106) | -1.21 (0.102) | -1.38 (0.104) | -1.07 (0.102)
Statistical Analysis 1: Comparison: Placebo vs GSK189075 50 mg vs GSK189075 100 mg vs GSK189075 250 mg vs GSK189075 500 mg vs GSK189075 1000 mg; Placebo, GSK189075 50 mg, GSK189075 100 mg, GSK189075 250 mg, GSK189075 500 mg, GSK189075 1000 mg; Test type: Other — Tukey's trend test for dose response: Change= Baseline+Treatment; p < 0.001, ANCOVA — Tukey's trend test adjusts for multiplicity with statistical significance based on p-value <0.05; Change= Baseline+Treatment
Statistical Analysis 2: Comparison: Placebo vs GSK189075 50 mg vs GSK189075 100 mg vs GSK189075 250 mg vs GSK189075 500 mg; Placebo, GSK189075 50 mg, GSK189075 100 mg, GSK189075 250 mg, GSK189075 500 mg; Test type: Other — Tukey's trend test for dose response; p < 0.001, ANCOVA — Tukey's trend test adjusts for multiplicity with statistical significance based on p-value <0.05
Statistical Analysis 3: Comparison: Placebo vs GSK189075 50 mg vs GSK189075 100 mg vs GSK189075 250 mg; Placebo, GSK189075 50 mg, GSK189075 100 mg, GSK189075 250 mg; Test type: Other — Tukey's trend test for dose response; p < 0.001, ANCOVA — Tukey's trend test adjusts for multiplicity with statistical significance based on p-value <0.05; Change=Baseline+Treatment
Statistical Analysis 4: Comparison: Placebo vs GSK189075 50 mg vs GSK189075 100 mg; Placebo, GSK189075 50 mg, GSK189075 100 mg; Test type: Other — Tukey's trend test for dose response; p < 0.001, ANCOVA — Tukey's trend test adjusts for multiplicity with statistical significance based on p-value <0.05; Change=Baseline+Treatment
Statistical Analysis 5: Comparison: Placebo vs GSK189075 50 mg; Placebo, GSK189075 50 mg; Test type: Other — Tukey's trend test for dose response; p < 0.001, ANCOVA — Tukey's trend test adjusts for multiplicity with statistical significance based on p-value <0.05; Change=Baseline+Treatment
Statistical Analysis 6: Comparison: Placebo vs GSK189075 50 mg; Placebo vs. GSK189075 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison included for informational purposes and not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -0.73, 95% CI 2-sided [-1.02 to -0.44]
Statistical Analysis 7: Comparison: Placebo vs GSK189075 100 mg; Placebo vs. GSK189075 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison included for informational purposes and not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -0.64, 95% CI 2-sided [-0.94 to -0.35]
Statistical Analysis 8: Comparison: Placebo vs GSK189075 250 mg; Placebo vs. GSK189075 250 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison included for informational purposes and not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -0.74, 95% CI 2-sided [-1.03 to -0.44]
Statistical Analysis 9: Comparison: Placebo vs GSK189075 500 mg; Placebo vs. GSK189075 500 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison included for informational purposes and not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -0.90, 95% CI 2-sided [-1.19 to -0.61]
Statistical Analysis 10: Comparison: Placebo vs GSK189075 1000 mg; Placebo vs. GSK189075 1000 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison included for informational purposes and not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -1.07, 95% CI 2-sided [-1.36 to -0.77]
Statistical Analysis 11: Comparison: Placebo vs Pioglitazone 30 mg; Placebo vs. Pioglitazone 30 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison included for informational purposes and not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -0.76, 95% CI 2-sided [-1.05 to -0.47]

2. Secondary Outcome: Change From Baseline in HbA1c (%) at Weeks 4 and 8
Description: Fasted blood samples for HbA1c were collected at Baseline and Weeks 4 and 8. Participants were required to fast for at least 8 hours prior to laboratory samples and were told not to take the morning dose of study medication on these visit days and to refrain from eating until instructed to do so by study personnel in the clinic. When the participant had not fasted, the participant was rescheduled to return to the clinic to have a fasted sample taken. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 4 and Week 8
Population: ITT Population with LOCF. Only those participants with a value at Baseline and at specified visits (after LOCF) were used for this analysis. One extreme outlier participant had withdrawn from Placebo arm due to lack of efficacy.
Measure: Mean (Standard Deviation); unit: Percentage of hemoglobin
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 47 | 46 | 44 | 45 | 47 | 47 | 47
Percentage of hemoglobin
  Week 4: number analyzed (Participants) | 41 | 45 | 42 | 44 | 45 | 45 | 46
  Week 4 | -0.30 (0.535) | -0.77 (0.541) | -0.69 (0.583) | -0.64 (0.535) | -0.83 (0.639) | -0.84 (0.551) | -0.39 (0.557)
  Week 8: number analyzed (Participants) | 43 | 45 | 43 | 44 | 47 | 45 | 47
  Week 8 | -0.41 (0.689) | -0.98 (0.712) | -0.96 (0.827) | -0.99 (0.751) | -1.07 (0.747) | -1.28 (0.636) | -0.88 (0.713)

3. Secondary Outcome: Change From Baseline to Week 12 in Fasting Plasma Glucose (FPG) at Weeks 4, 8 and 12
Description: Fasted blood samples for FPG were collected up to Week 12. Participants were required to fast for at least 8 hours prior to laboratory samples and were told not to take the morning dose of study medication on these visit days and to refrain from eating until instructed to do so by study personnel in the clinic. When the participant had not fasted, the participant was rescheduled to return to the clinic to have a fasted sample taken. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 4, Week 8 and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 46 | 46 | 44 | 43 | 46 | 46 | 46
Millimoles per Liter (mmol/L)
  Week 4 | -0.49 (1.991) | -0.56 (1.512) | -1.43 (2.005) | -1.49 (2.314) | -1.90 (2.232) | -2.48 (2.491) | -1.26 (1.294)
  Week 8 | -0.62 (1.859) | -0.91 (2.073) | -1.30 (1.821) | -1.76 (2.137) | -2.14 (2.547) | -2.78 (2.531) | -1.73 (1.340)
  Week 12 | -0.51 (1.700) | -0.89 (1.960) | -1.63 (2.145) | -1.80 (2.107) | -2.07 (2.459) | -2.76 (2.821) | -1.71 (1.978)

4. Secondary Outcome: Change From Baseline to Week 12 in Fructosamine
Description: Fasted blood samples for fructosamine were collected up to Week 12. Participants were required to fast for at least 8 hours prior to laboratory samples and were told not to take the morning dose of study medication on these visit days and to refrain from eating until instructed to do so by study personnel in the clinic. When the participant had not fasted, the participant was rescheduled to return to the clinic to have a fasted sample taken. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) to Week 12
Population: ITT Population with LOCF. Only those participants with a value at Baseline up to Week 12 (after LOCF) were used for this analysis.
Measure: Mean (Standard Deviation); unit: Micromol per Liter (mcmol/L)
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 39 | 37 | 37 | 36 | 41 | 39 | 43
Micromol per Liter (mcmol/L) | 5.7 (51.24) | -33.8 (38.20) | -35.7 (41.69) | -38.9 (29.62) | -41.9 (35.54) | -55.2 (30.31) | -34.7 (38.84)

5. Secondary Outcome: Change From Baseline to Week 12 in Fasting Insulin
Description: Fasted blood samples for insulin were collected up to Week 12. Participants were required to fast for at least 8 hours prior to laboratory samples and were told not to take the morning dose of study medication on these visit days and to refrain from eating until instructed to do so by study personnel in the clinic. When the participant had not fasted, the participant was rescheduled to return to the clinic to have a fasted sample taken. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) to Week 12
Population: ITT Population with LOCF. Only those participants with a value at Baseline and up to Week 12 (after LOCF) were used for this analysis.
Measure: Mean (Standard Deviation); unit: Picomol per Liter (pmol/L)
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 38 | 40 | 40 | 39 | 41 | 43 | 42
Picomol per Liter (pmol/L) | -30.6 (171.35) | 0.3 (58.69) | -20.7 (60.75) | -9.7 (43.95) | -25.8 (60.94) | -15.1 (57.59) | -2.1 (49.60)

6. Secondary Outcome: Number of Participants at Week 12 With: HbA1c <= 6.5%, HbA1c <7.0%; FPG <7 Mmo/L, FPG <7.8 mmol/L; FPG <5.5 mmol/L; a Decrease From Baseline of HbA1c >= 0.7%; a Decrease From Baseline of FPG ≥1.7 mmol/L
Description: Fasted blood samples for HbA1c were collected at Week 12. Participants were required to fast for at least 8 hours prior to laboratory samples and were told not to take the morning dose of study medication on these visit days and to refrain from eating until instructed to do so by study personnel in the clinic. When the participant had not fasted, the participant was rescheduled to return to the clinic to have a fasted sample taken. Number of participants at Week 12 with: HbA1c <= 6.5%, HbA1c <7.0%; FPG <7 mmo/L (126 milligram/deciliter [mg/dL]), FPG <7.8 mmol/L (140 mg/dL); FPG <5.5 mmol/L (100 mg/dL); a decrease from Baseline of HbA1c >= 0.7%; a decrease from Baseline of FPG ≥1.7 mmol/L (30 mg/dL) are presented.
Time Frame: Week 12
Population: ITT Population with Last Observation Carried Forward (LOCF). Only those participants with a value at Baseline and at Week 12 (after LOCF) were used for this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 47 | 46 | 44 | 45 | 47 | 47 | 47
Participants
  HbA1c <= 6.5%: number analyzed (Participants) | 44 | 45 | 43 | 44 | 47 | 45 | 47
  HbA1c <= 6.5% | 3 | 10 | 8 | 11 | 17 | 17 | 8
  HbA1c <7.0%: number analyzed (Participants) | 44 | 45 | 43 | 44 | 47 | 45 | 47
  HbA1c <7.0% | 9 | 20 | 18 | 22 | 28 | 29 | 21
  FPG <7 mmo/L: number analyzed (Participants) | 47 | 46 | 44 | 43 | 46 | 46 | 46
  FPG <7 mmo/L | 4 | 16 | 20 | 18 | 22 | 22 | 21
  FPG <7.8 mmol/L: number analyzed (Participants) | 47 | 46 | 44 | 43 | 46 | 46 | 46
  FPG <7.8 mmol/L | 13 | 24 | 26 | 27 | 33 | 34 | 31
  FPG <5.5 mmol/L: number analyzed (Participants) | 47 | 46 | 44 | 43 | 46 | 46 | 46
  FPG <5.5 mmol/L | 0 | 4 | 2 | 5 | 4 | 3 | 2
  Decrease from Baseline of HbA1c >= 0.7%: number analyzed (Participants) | 44 | 45 | 43 | 44 | 47 | 45 | 47
  Decrease from Baseline of HbA1c >= 0.7% | 16 | 33 | 27 | 33 | 36 | 39 | 28
  Decrease from Baseline of FPG ≥1.7 mmol/L: number analyzed (Participants) | 47 | 46 | 44 | 43 | 46 | 46 | 46
  Decrease from Baseline of FPG ≥1.7 mmol/L | 8 | 15 | 19 | 21 | 24 | 30 | 23

7. Secondary Outcome: Percent Change From Baseline in Lipid Parameters at Weeks 4, 8 and 12(Triglycerides [TG], Total Cholesterol [TC], Low-density Lipoprotein Cholesterol [LDL-C] and High-density Lipoprotein Cholesterol [HDL-C])
Description: Fasted samples for TC, LDL-C, HDL-C and TG were collected at Week 12. When the participant had not fasted, the participant was rescheduled to return to the clinic to have a fasted sample taken. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. Percent Change based on log-transformed data: 100*(exponentiated(mean change on log scale)-1)
Time Frame: Baseline (Week 0) and Week 4, Week 8 and Week 12
Population: ITT Population with LOCF. Only those participants with a value at Baseline and at specified visits (after LOCF) were used for this analysis.
Measure: Median (Full Range); unit: Percent change
Groups:
- Pioglitazone 30mg: Eligible participants received Pioglitazone 30 mg tablets, orally, once daily before breakfast for 12 weeks.
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30mg
Number analyzed (Participants) | 47 | 46 | 44 | 45 | 47 | 47 | 47
Percent change
  TG: Week 4: number analyzed (Participants) | 44 | 45 | 42 | 44 | 44 | 46 | 46
  TG: Week 4 | -8.35 [-44.3 to 110.1] | -3.45 [-48.1 to 177.8] | 6.32 [-55.1 to 112.1] | -13.42 [-56.8 to 133.6] | -13.04 [-74.8 to 207.1] | -4.62 [-48.2 to 256.3] | -7.22 [-68.6 to 76.9]
  TG: Week 8: number analyzed (Participants) | 46 | 45 | 43 | 44 | 47 | 46 | 47
  TG: Week 8 | -1.66 [-67.2 to 135.2] | -9.09 [-61.3 to 88.8] | 0.59 [-47.4 to 122.5] | -10.01 [-57.9 to 100.0] | -13.35 [-51.9 to 207.1] | -7.30 [-60.9 to 121.6] | -0.79 [-71.1 to 82.5]
  TG: Week 12: number analyzed (Participants) | 46 | 45 | 43 | 44 | 47 | 46 | 47
  TG: Week 12 | 3.32 [-58.6 to 135.2] | -10.91 [-60.2 to 213.0] | 10.92 [-45.3 to 232.5] | -4.71 [-56.8 to 73.6] | -15.28 [-66.8 to 255.7] | -9.97 [-58.4 to 123.4] | -7.19 [-58.2 to 116.7]
  TC: Week 4: number analyzed (Participants) | 44 | 45 | 42 | 44 | 44 | 46 | 46
  TC: Week 4 | 0.47 [-57.4 to 25.8] | 1.85 [-22.9 to 65.0] | 1.62 [-17.6 to 34.8] | 4.13 [-40.1 to 63.9] | 4.43 [-37.9 to 36.6] | 2.39 [-22.7 to 54.4] | 2.29 [-42.0 to 29.5]
  TC: Week 8: number analyzed (Participants) | 46 | 45 | 43 | 44 | 47 | 46 | 47
  TC: Week 8 | 0.82 [-48.4 to 48.4] | 3.49 [-31.3 to 43.1] | 3.64 [-31.5 to 30.0] | 4.49 [-14.0 to 73.7] | 5.31 [-19.9 to 41.2] | 0.00 [-24.3 to 49.9] | 1.06 [-40.2 to 34.9]
  TC: Week 12: number analyzed (Participants) | 46 | 45 | 43 | 44 | 47 | 46 | 47
  TC: Week 12 | 4.75 [-46.5 to 76.6] | 3.39 [-28.1 to 43.4] | 5.45 [-19.0 to 84.6] | 3.97 [-16.8 to 67.1] | 9.82 [-16.3 to 43.3] | 2.77 [-17.5 to 52.5] | -2.05 [-48.3 to 31.4]
  LDL-C: Week 4: number analyzed (Participants) | 42 | 43 | 40 | 43 | 43 | 41 | 45
  LDL-C: Week 4 | 0.82 [-75.6 to 68.5] | 0.83 [-27.3 to 117.0] | 0.37 [-30.9 to 75.0] | 6.91 [-52.9 to 84.1] | 10.03 [-39.0 to 59.6] | 7.02 [-37.0 to 130.3] | 0.00 [-54.0 to 50.0]
  LDL-C: Week 8: number analyzed (Participants) | 45 | 44 | 42 | 43 | 46 | 44 | 46
  LDL-C: Week 8 | 3.17 [-63.0 to 56.4] | 8.67 [-38.7 to 53.1] | 3.62 [-32.6 to 125.0] | 8.96 [-37.9 to 118.8] | 7.57 [-24.8 to 67.2] | 4.44 [-39.5 to 119.5] | -2.24 [-47.8 to 55.2]
  LDL-C: Week 12: number analyzed (Participants) | 45 | 44 | 43 | 44 | 47 | 44 | 46
  LDL-C: Week 12 | 3.17 [-60.4 to 56.4] | 6.69 [-39.4 to 90.2] | 3.57 [-29.7 to 355.0] | 3.93 [-23.0 to 102.9] | 11.43 [-36.7 to 92.0] | 14.89 [-23.7 to 125.6] | 1.18 [-61.9 to 51.8]
  HDL-C: Week 4: number analyzed (Participants) | 44 | 45 | 42 | 44 | 44 | 46 | 46
  HDL-C: Week 4 | -1.97 [-23.5 to 23.5] | 5.43 [-11.5 to 45.8] | 3.69 [-31.3 to 54.2] | 5.13 [-29.3 to 93.3] | 5.69 [-17.0 to 56.2] | 0.00 [-33.0 to 32.9] | 9.18 [-17.6 to 57.5]
  HDL-C: Week 8: number analyzed (Participants) | 46 | 45 | 43 | 44 | 47 | 46 | 47
  HDL-C: Week 8 | 0.00 [-31.6 to 19.1] | 6.20 [-20.6 to 40.6] | 5.00 [-20.7 to 58.3] | 3.09 [-41.4 to 93.5] | 7.14 [-15.8 to 59.2] | 0.00 [-42.7 to 52.2] | 8.20 [-13.2 to 48.1]
  HDL-C: Week 12: number analyzed (Participants) | 46 | 45 | 43 | 44 | 47 | 46 | 47
  HDL-C: Week 12 | 0.00 [-31.6 to 32.6] | 5.56 [-28.6 to 42.2] | 4.96 [-16.7 to 70.8] | 6.70 [-14.4 to 90.3] | 11.93 [-15.8 to 51.7] | 4.27 [-50.2 to 36.4] | 10.00 [-12.6 to 46.2]

8. Secondary Outcome: Change From Baseline to Week 12 in Body Weight
Description: Weight of participants was measured from Baseline (Week 0) to Week 12 and recorded in the case report form (CRF). Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) to Week 12
Population: ITT population with LOCF for withdrawn participants or missing values.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 47 | 46 | 44 | 45 | 47 | 47 | 47
Kilograms | -0.49 (1.719) | -1.78 (3.197) | -2.41 (2.850) | -2.38 (2.875) | -3.52 (2.874) | -4.00 (2.945) | 0.96 (2.425)

9. Secondary Outcome: Change From Baseline to Week 12 in Waist Circumference
Description: Waist circumference of participants was measured from Baseline (Week 0) to Week 12 and recorded in the CRF. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) to Week 12
Population: ITT population with LOCF for withdrawn participants or missing values.
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 41 | 43 | 43 | 43 | 42 | 44 | 47
Centimeters | -0.7 (2.92) | -1.2 (3.58) | -2.0 (4.51) | -2.2 (3.43) | -2.6 (3.31) | -2.4 (4.26) | 1.3 (4.82)

10. Secondary Outcome: Change From Baseline in 24-hour Percent of Filtered Glucose Excreted in Urine
Description: A 24-hour urine collection was obtained from all participants at Baseline (Week 0) and Week 12 to measure glucose. Participants were provided with urine collection bottles and cooler prior to these visits and instructed that the urine collections must be kept cold and dropped off at the clinic prior to or at the scheduled visits. Site staff queried participants to determine whether the sample represented a full 24-hour collection. The total volume and the sample date and time were recorded. The entire 24-hour urine collection was well mixed in one container and a urine aliquot obtained. Samples were assayed for glucose. The 24-hour collections were used to derive 24-hour urine glucose excretion corrected for filtered load. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12 (24-hour urine collection)
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of filtered glucose molecules
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 23 | 28 | 27 | 27 | 25 | 27 | 37
Percentage of filtered glucose molecules | -1.09 (5.731) | 27.96 (15.693) | 40.43 (16.144) | 38.98 (19.006) | 42.41 (22.708) | 52.39 (15.264) | -0.99 (2.313)

11. Secondary Outcome: Change From Baseline in Plasma Glucose Area Under the Curve (AUC) During a 2-hour Oral Glucose Tolerance Test (OGTT)
Description: Post-prandial assessments of glucose were performed at Baseline (Week 0) and at Week 12 using a 2-hour OGTT in a subgroup of participants at selected sites who agreed to participate. Participants were required to fast for at least 8 hours prior to the test. Seventy-five (75) g of standard oral glucose solution was administered 15 minutes after the morning administration of study medication (Week 12) and in the place of breakfast at Week 0 (i.e., at Week 0 the OGTT was completed prior to administration of study medication). Time "0" started when the participants drank the glucose solution. Blood samples were collected at the following times relative to the administration of oral glucose: -30 min (pre-glucose), -20 min (pre-glucose), 20 min, 30 min, 1 hour, 1.5 hour and 2 hour post glucose administration. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12 (0 to 2 hour OGTT)
Population: The OGTT Population with LOCF which comprised of participants in the ITT population having evaluable Baseline and corresponding on-therapy OGTT measurements (for at least one of the measured parameters of FPG, C-Peptide or Insulin). Only those participants with a value at Baseline and at Week 12 (after LOCF) were used for this analysis.
Measure: Mean (Standard Deviation); unit: Millimol*hour per Liter (mmol*hr/L)
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 9 | 8 | 12 | 8 | 10 | 14 | 7
Millimol*hour per Liter (mmol*hr/L) | -0.90 (5.739) | -6.31 (5.907) | -6.71 (7.326) | -7.69 (3.791) | -6.06 (2.837) | -7.59 (3.065) | -6.55 (3.841)

12. Secondary Outcome: Change From Baseline in Insulin AUC During a 2-hour OGTT
Description: Post-prandial assessments of insulin were performed at Baseline (Week 0) and at Week 12 using a 2-hour OGTT in a subgroup of participants at selected sites who agreed to participate. Participants were required to fast for at least 8 hours prior to the test. Seventy-five (75) g of standard oral glucose solution was administered 15 minutes after the morning administration of study medication (Week 12) and in the place of breakfast at Week 0 (i.e., at Week 0 the OGTT was completed prior to administration of study medication). Time "0" started when the participants drank the glucose solution. Blood samples were collected at the following times relative to the administration of oral glucose: -30 min (pre-glucose), -20 min (pre-glucose), 20 min, 30 min, 1 hour, 1.5 hour and 2 hour post glucose administration. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12 (0 to 2-hour OGTT)
Population: OGTT with LOCF Population. Only those participants with a value at Baseline and at Week 12 (after LOCF) were used for this analysis.
Measure: Mean (Standard Deviation); unit: Picomol*hour per Liter (pmol*hr/L)
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 8 | 8 | 12 | 8 | 9 | 13 | 9
Picomol*hour per Liter (pmol*hr/L) | -5.3 (177.23) | 162.4 (362.82) | -70.9 (193.77) | 66.6 (213.07) | -173.9 (143.52) | -97.8 (224.24) | 10.0 (128.77)

13. Secondary Outcome: Change From Baseline in C-peptide AUC During a 2-hr OGTT
Description: Post-prandial assessments of C-peptide were performed at Baseline (Week 0) and at Week 12 using a 2-hour OGTT in a subgroup of participants at selected sites who agreed to participate. Participants were required to fast for at least 8 hours prior to the test. Seventy-five (75) g of standard oral glucose solution was administered 15 minutes after the morning administration of study medication (Week 12) and in the place of breakfast at Week 0 (i.e., at Week 0 the OGTT was completed prior to administration of study medication). Time "0" started when the participants drank the glucose solution. Blood samples were collected at the following times relative to the administration of oral glucose: -30 min (pre-glucose), -20 min (pre-glucose), 20 min, 30 min, 1 hour, 1.5 hour and 2 hour post glucose administration. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12 (0 to 2 hour OGTT)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Nanomol*hour per Liter (nmol*hr/L)
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 8 | 8 | 12 | 7 | 9 | 12 | 9
Nanomol*hour per Liter (nmol*hr/L) | -0.140 (0.7348) | 0.654 (1.4023) | -0.156 (1.0566) | -0.026 (0.9606) | -0.476 (0.4668) | -0.175 (0.8322) | -0.239 (0.6732)

14. Secondary Outcome: Number of Participants With On-therapy Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
Time Frame: Up to 12 weeks
Population: Safety population which comprised of all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 48 | 47 | 48 | 48 | 48 | 47 | 48
Participants
  AE | 18 | 18 | 17 | 19 | 18 | 22 | 22
  SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With On-therapy Hypoglycemia
Description: Hypoglycemia is low blood glucose or low blood sugar. Hypoglycemic events were collected separately and reported separately from AE, including supplemental data which were not collected for AE. However, any hypoglycemic event which met the criteria for a SAE was included in the SAE summaries. The number of participants in each group that experienced a hypoglycemic event was summarized by frequency of the events.
Time Frame: Up to 14 weeks
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 48 | 47 | 48 | 48 | 48 | 47 | 48
Participants | 1 | 1 | 0 | 0 | 1 | 0 | 0

16. Secondary Outcome: Number of Participants With Change From Baseline Vital Signs of Potential Clinical Concern
Description: Vital signs included heart rate and blood pressure. Heart rate and blood pressure were taken before blood draws were performed. Participants were asked to refrain from smoking for at least 30 minutes prior to vital sign measurements. Heart rate and blood pressure was measured pre-dose in duplicate at the specified visits, after the participant had been lying quietly for 5 minutes, and then in duplicate 3 minutes after standing up. Heart rate was measured at the same time as blood pressure using the standardized blood pressure equipment that was provided. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Up to 14 weeks
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 48 | 47 | 48 | 48 | 48 | 47 | 48
Participants
  High SBP: number analyzed (Participants) | 47 | 46 | 44 | 45 | 47 | 47 | 47
  High SBP | 3 | 0 | 2 | 0 | 0 | 1 | 0
  Low SBP: number analyzed (Participants) | 47 | 46 | 44 | 45 | 47 | 47 | 47
  Low SBP | 0 | 0 | 1 | 2 | 2 | 2 | 0
  High DBP: number analyzed (Participants) | 47 | 46 | 44 | 45 | 47 | 47 | 47
  High DBP | 1 | 0 | 0 | 0 | 0 | 2 | 0
  Low DBP: number analyzed (Participants) | 47 | 46 | 44 | 45 | 47 | 47 | 47
  Low DBP | 0 | 1 | 2 | 0 | 0 | 1 | 3
  High heart rate: number analyzed (Participants) | 47 | 46 | 44 | 45 | 47 | 47 | 47
  High heart rate | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Low heart rate: number analyzed (Participants) | 47 | 46 | 44 | 45 | 47 | 47 | 47
  Low heart rate | 0 | 0 | 0 | 0 | 1 | 1 | 0

17. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Values of Potential Clinical Concern
Description: Full 12-lead ECGs were recorded at screening, Baseline (Week 0), Week 4, Week 12 or early withdrawal, and Week 14 (Follow-up) using an ECG machine that automatically calculated the heart rate and measured the PR, QRS, QT and corrected QT (QTc) intervals. All 12-lead ECGs were read locally by the Investigator or his/her designate and were forwarded electronically to the central reader for interpretation. If the QTc was >500 milliseconds (msec) on the locally read ECG recording, an additional 2 ECG recordings at 10 minute intervals were made at that visit. If the average QTc for the 3 recordings was >500 msec, the participant was withdrawn from the study.
Time Frame: Up to Early withdrawal (Between Week 12 and Week 14)
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 46 | 45 | 43 | 44 | 47 | 46 | 47
Participants
  PR interval > 300 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS Duration > 200 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTc(Bazett) > 500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTc(Fridericia) > 500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Change From Baseline in Standard Laboratory Parameters of Potential Clinical Concern
Description: Participants were instructed to fast for at least 8 hours prior to all study visits for the collection of laboratory samples. An additional fasting blood sample (serum and plasma) was drawn at Week 0, Week 4, Week 6 and Week 12 or at early withdrawal (up to 14 weeks) and kept in long-term storage for future testing of biomarkers for diabetes and complications of the disease. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Up to 14 weeks
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
Number analyzed (Participants) | 46 | 46 | 44 | 44 | 47 | 46 | 47
Participants
  Low Hemoglobin | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Low Hematocrit | 1 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 weeks.
Description: On-therapy SAE and non-SAEs are reported for the Safety population which comprised of all participants who received at least one dose of study medication.
Arm/Group | Placebo | GSK189075 50 mg | GSK189075 100 mg | GSK189075 250 mg | GSK189075 500 mg | GSK189075 1000 mg | Pioglitazone 30 mg
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47 | 0/48 | 0/48 | 0/48 | 0/47 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/47 | 0/48 | 0/48 | 0/48 | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 3/48 | 5/47 | 5/48 | 4/48 | 5/48 | 3/47 | 12/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | GSK189075 50 mg (N=47) | GSK189075 100 mg (N=48) | GSK189075 250 mg (N=48) | GSK189075 500 mg (N=48) | GSK189075 1000 mg (N=47) | Pioglitazone 30 mg (N=48)
Headache (Nervous system disorders) | 0 | 1 | 2 | 1 | 2 | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 0 | 2 | 3
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.